CLINICAL TRIAL: NCT03804736
Title: Fecal Microbiota Transplant by Oral Capsules Enriched With Lactobacilli for Recurrent Clostridium Difficile Infection
Brief Title: Fecal Microbiota Transplant by Oral Capsules With Lactobacilli for Recurrent Clostridium Difficile Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Adrián Camacho-Ortiz, Principal Investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IF-0016-3
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-03

CONDITIONS: Clostridium Difficile Infection
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients were randomized by a closed envelope method in a 1: 1 ratio to either FMT-c (15 capsules every 12 h by 2 days) or a FMT-c and Lactobacillus (15 capsules every 12 h by 2 days)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FMT-c (Active Comparator): Patients in this arm received FMT-c (15 capsules every 12 h for 2 days)
  Interventions: Biological: FMT-c
- FMT-c lactobacillus (Experimental): Patients in this arm received FMT-c Lactobacillus (15 capsules every 12 h for 2 days)
  Interventions: Biological: FMT-c Lactobacillus

INTERVENTIONS:
Biological: FMT-c — Patients in the FMT-c receive FMT-c (15 capsules every 12 h for 2 days)
  Arms: FMT-c
Biological: FMT-c Lactobacillus — Patients in the FMT-c Lactobacillus receive FMT-c Lactobacillus (15 capsules every 12 h for 2 days)
  Arms: FMT-c lactobacillus

SUMMARY:
Investigators designed an open, two-arm study to compare fecal microbiota transplant by oral capsules (FMT-c ) versus FMT-c enriched with Lactobacillus for treatment of C. difficile recurrent infection

DETAILED DESCRIPTION:
Investigators designed an open, two-arm study to compare to compare fecal microbiota transplant by oral capsules (FMT-c ) versus FMT-c enriched with Lactobacillus for treatment of C. difficile recurrent infection.

From each patient, a fecal sample was obtained at days 0, 3, and 7 after treatment. Fecal samples are analyzed by 16 subunit ribosomal ribonucleic acid (16S rRNA) metagenomic sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years With recurrent CDI

Exclusion Criteria:Older than 18 years

-

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-11-01; Primary Completion 2018-06-30 (Actual); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
decrease in the number of evacuations | up to two days
  The cure of CDI was measured